CLINICAL TRIAL: NCT04306627
Title: Evaluation of Carotid Intima Media Thickness by Treatment of Vascular and Metabolic Factors With Combined Antihypertensive and Hypolipidemic Therapy
Brief Title: Effect of Atorvastatin on Carotid Intima Media Thickness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yerevan State Medical University (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YerevanStateMU
Record Dates: First submitted 2020-02-24; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Essential Hypertension; Hypercholesterolemia
Keywords: arterial hypertension; statin; carotid artery intima-media thickness
MeSH Terms: conditions — Essential Hypertension; Hypercholesterolemia; Hypertension | interventions — Perindopril; Amlodipine

STUDY DESIGN:
Intervention Model Description: Endpoints of study The primary endpoints in the study is the change in mean IMT of the CCA from baseline to 6 months in two groups and antihypertensive treatment efficacy in both groups .
  The secondary endpoints are assessment of level of total and LDL cholesterol concentrations in blood plasma after 6 months of treatment in both groups and correlation between carotid IMT and values of total cholesterol and LDL levels in blood plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perindopril/Amlodipine arm (Active Comparator): Patients will be preliminary screened before 7-10 days for clinical and laboratory examination to meet eligibility criteria for inclusion in study.
  Perindopril+amlodipine combination doses will be up titrated over two weeks in case of need to control adequate arterial blood pressure < 140/90. The 4 doses combinations and their adjustments will be made by investigating physician according to guideline based treatment of arterial hypertension and dyslipidemia.
  Interventions: Drug: Perindopril/Amlodipine and Perindopril/Amlodipine/Atorvastatin treatment
- Perindopril/Amlodipine/Atorvastatin arm (Active Comparator): Subjects should not previously be on statin therapy and subjects who needs to be will start atorvastatin in combination treatment pill . We will study the effects of 6-month treatment with perindopril +amlodipin+atorvastatin combination on plasma concentrations of total cholesterol and LDL cholesterol.
  Interventions: Drug: Perindopril/Amlodipine and Perindopril/Amlodipine/Atorvastatin treatment

INTERVENTIONS:
Drug: Perindopril/Amlodipine and Perindopril/Amlodipine/Atorvastatin treatment — comparative antihypertensive antilipidemic treatment assessment on carotid intima media thickness in both study groups

SUMMARY:
The investigators hypothesize that additive effects of combined antihypertensive medications and statin in a single pill combination may better reduce progression of vascular remodeling and inhibit atherosclerosis progression. The fixed association of atorvastatin, perindopril and amlodipine under the name of Lipertance is the first fixed combination of these three groups to control the risk factors that are hypertension and dyslipidemia which can be used both in primary and secondary cardiovascular prevention .

DETAILED DESCRIPTION:
Eligible participants with appropriately signed informed consent will be randomized to either the perindopril+amlodipin or perindopril+amlodipin+atorvastatin combinations.

Patients will be preliminary screened before 7-10 days for clinical and laboratory examination to meet eligibility criteria for inclusion in study.

Perindopril+amlodipine combination doses will be up titrated over two weeks in case of need to control adequate arterial blood pressure < 140/90. The 4 doses combinations and their adjustments will be made by investigating physician according to guideline based treatment of arterial hypertension and dyslipidemia.

Subjects should not previously be on statin therapy and subjects who needs to be will start atorvastatin in combination treatment pill . The investigators will study the effects of 6-month treatment with perindopril +amlodipin+atorvastatin combination on plasma concentrations of total cholesterol and LDL cholesterol. Liver enzyme markers will be assessed in patients on additional statin treatment on day 90 for safety assessment. All participants will be followed-up for 6 months.

Inclusion criteria

* Patients aged between 45 and 85 years
* blood pressure ≥ 140/90 mmHg with one antihypertensive drug or 150/100 mHg for untreated patients
* plasma LDL-cholesterol concentrations > 2,5mm/L (without concomitant hypolipidemic drugs)
* at least one additional cardiovascular risk factor apart of arterial hypertension
* minimal thickness of intima media complex at least 0,8 mm.

Exclusion criteria

* premenopausal females with potential for pregnancy
* angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker therapy in the previous 3 months,
* initiation or change in dose of statin therapy within previous 3 months
* anticipated change in lipid lowering therapy
* acute coronary or cerebrovascular event within 2 months
* glomerular filtration rate < 30 ml/min
* previous history of side effects to RAAS inhibitors and Ca channel blocking agents
* inability to give informed consent
* inability to undergo carotid ultrasound examination.

Adverse events (AE)

Based on the intention-to-treat the patient population, safety will be checked by recording adverse effects throughout the study: severe AEs regardless as to whether or not there is causal relationship between the AEs and the study; and relevant AEs such as myalgia, cough , palpitations, peripheric edemas, diziness symptoms. When the investigators confirm these AEs, the grade of severity, procedures, outcomes, and relationship to the study drug will be assessed and recorded.

Serious adverse event (SAE)

A serious adverse event is an AE occurring during any study phase and at any dose of the investigational product that fulfills one or more of the following criteria: results in death, is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above.

The Investigator must inform the Sponsor of any SAE that occurs in the course of the study within 48 hours of when he or she becomes aware of it.

Carotid Ultrasound An ultrasound linear probe with 5-10 MHz linear transducer will be used for measuring the carotid artery intima media thickness ( IMT ). The carotid artery will be scanned by 3 trained in vascular ultrasound and echocardiography physicians. All study subjects will be examined in the supine position with the head tilted backward. Measurements of the left and right IMT of the posterior wall of the common carotid, 1 cm distal to the bulb bifurcation, by ultrasound 2D exam will be performed

Blood pressure (BP) will be measured at the University Cardiology Clinic by a trained nurse or physician using a calibrated and validated digital sphygmomanometer. BP measurements will be taken with the patient in a seated position with the arm supported at heart level, after a 5 min rest and after abstaining from food, beverages containing caffeine, and smoking for at least 2 h prior to BP measurement. BP will be recorded as three serial measurements at intervals of 30 sec on both arms.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged between 45 and 85 years

  * blood pressure ≥ 140/90 mmHg with one antihypertensive drug or 150/100 mHg for untreated patients
  * plasma LDL-cholesterol concentrations > 4.1 mmol/L without hypolipidemic drugs within the last 6 months
  * at least one additional cardiovascular risk factor apart of arterial hypertension
  * minimal thickness of intima media complex at least 0,8 mm.

Exclusion Criteria:

* premenopausal females with potential for pregnancy
* angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker therapy in the previous 3 months,
* initiation or change in dose of statin therapy within previous 3 months
* anticipated change in lipid lowering therapy
* acute coronary or cerebrovascular event within 2 months
* glomerular filtration rate < 30 ml/min
* previous history of side effects to RAAS inhibitors and Ca channel blocking agents
* inability to give informed consent
* inability to undergo carotid ultrasound examination

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-10-16 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
The change in mean IMT of the CCA from baseline to 6 months in two groups and antihypertensive treatment efficacy in both groups . | 6 months
  The fixed association of atorvastatin, perindopril and amlodipine is the first fixed combination of these three groups to control the risk factors that are hypertension and dyslipidemia. Additive effects of combined antihypertensive medications and statin in a single pill combination may better reduce progression of vascular remodeling and inhibit atherosclerosis progression.

SECONDARY OUTCOMES:
Assessment of level of total and LDL cholesterol concentrations in blood plasma after 6 months of treatment in both groups. | 6 months
  Assessment of level of total and LDL cholesterol concentrations in blood plasma after 6 months of treatment in both groups and correlation between carotid IMT and values of total cholesterol and LDL levels in blood plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Hamayak Sisakian, MD, Principal Investigator — Yerevan State Medical University

IPD SHARING:
Plan to Share IPD: No